CLINICAL TRIAL: NCT00231959
Title: A Double-Blind Placebo-Controlled Trial of Adjunctive Pramipexole, a Dopamine Receptor Agonist, for Treatment Resistant Major Depressive Episodes
Brief Title: Effectiveness of Pramipexole for Treatment-Resistant Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Roy Perlis, Director, Center for Experimental Drugs and Diagnostics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23MH067060 (NIH); K23MH067060 (NIH); DATR AK-TNGP1
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Depression
Keywords: Depression, Treatment-Resistant
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Pramipexole (Experimental)
  Interventions: Drug: Pramipexole (Mirapex)

INTERVENTIONS:
Drug: Pramipexole (Mirapex) — pramipexole 0.5mg tablets qd and titrated per protocol
  Arms: Pramipexole
Drug: Placebo — sugar pill
  Arms: Sugar pill

SUMMARY:
This study will evaluate the effectiveness of pramipexole (Mirapex) in managing treatment-resistant depression.

DETAILED DESCRIPTION:
Depression is a serious medical illness, for which various types of treatment have been developed. Both medications and therapies have proven effective in treating depression. However, some people with depression do not benefit from these treatments. New medications are needed for treating depression in those who have not responded to commonly used antidepressants. Pramipexole (Mirapex) is most often used for the treatment of Parkinson's disease, but has been reported to have antidepressant effects as well. This study will evaluate the effectiveness of pramipexole in treating depression in individuals that have not responded to other medications.

Participants in this double blind study will be randomly assigned to receive either pramipexole or placebo, in addition to their current medications, for 8 weeks. Treatment response will be assessed at the end of this phase by measuring symptoms of depression. At this time, those individuals who have responded to treatment will have the option to continue in a 6-month follow-up study. Participants will be seen monthly throughout the 6 months to assess treatment response. Participants who do not exhibit a response to treatment will be tapered off the medication. All participants will receive 3 months of follow-up care, regardless of their response to the medication.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for major depressive disorder
* Meets criteria for current major depressive episode
* Score of at least 18 on the Montgomery-Asberg Depression Rating Scale (MADRS) at the baseline visit
* Currently being treated with antidepressant monotherapy at an adequate dose for 6 weeks or willing to enter open lead-in treatment
* Agrees to use an effective form of contraception throughout the study

Exclusion Criteria:

* Pregnant
* At risk for suicide or homicide
* Unstable medical illness (e.g., cardiovascular, liver, kidney, respiratory, endocrine, or neurologic disease, including uncontrolled seizure disorder)
* History of a substance use disorder within 6 months of study enrollment
* History of or current psychotic features
* Currently being treated with typical or atypical antipsychotic medications
* Currently being treated with a medication known to significantly decrease pramipexole clearance (e.g., cimetidine, ranitidine, diltazem, verapamil, quinine or triamterene)
* Clinical or laboratory evidence of untreated hypothyroidism
* History of a 2-week or longer course of pramipexole
* Intolerance of pramipexole at any dose
* Any investigational psychotropic drug use within the last three months
* Level 3 or greater antidepressant resistance as assessed by the ATHF
* Three or more episodes of self-harm in the year prior to study enrollment
* Documented history of poor treatment adherence or frequently missed appointments
* Parkinson's disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2003-09; Primary Completion 2007-09 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Score on the Montgomery-Asberg Depression Rating Scale | Measured at Week 8 and monthly for the duration of the 6-month optional continuation phase for responders
Clinical Global Impressions (CGI) scale | Measured at Week 8 and monthly for the duration of the 6-month optional continuation phase for responders

CONTACTS AND LOCATIONS:
Overall Officials: Roy Perlis, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Cusin C, Iovieno N, Iosifescu DV, Nierenberg AA, Fava M, Rush AJ, Perlis RH. A randomized, double-blind, placebo-controlled trial of pramipexole augmentation in treatment-resistant major depressive disorder. J Clin Psychiatry. 2013 Jul;74(7):e636-41. doi: 10.4088/JCP.12m08093. PMID 23945458